CLINICAL TRIAL: NCT05362981
Title: Contra-attitudinal Versus Mindfulness Treatment in Anorexia Nervosa - Randomised Controlled Trial
Brief Title: Contra-attitudinal Versus Mindfulness Treatment in Anorexia Nervosa Controlled Trial
Acronym: CAT-AN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2020-A02346-33
Record Dates: First submitted 2022-05-02; First posted 2022-05-05 (Actual); Last update posted 2023-06-09 (Actual); Status verified 2023-04

CONDITIONS: Anorexia Nervosa
MeSH Terms: conditions — Anorexia Nervosa

STUDY DESIGN:
Intervention Model Description: The patients will be recruited from the active files of the four centers participating in the study. In order to avoid the disappointment bias, they will be randomized into three groups, according to a procedure adapted from the Zelen method, in two stages. After verification of the inclusion criteria, eligible patients will receive initial information detailing the follow-up methods, but not the intervention. If patients agree to participate, they will be randomized to three groups: CAT, MBCT or usual management. Patients in the CAT and MBCT groups will then be informed of the group in which they have been randomized, will sign a new consent form and the corresponding intervention will be offered to them.
Masking Description: The patients will be recruited from the active files of the four centers participating in the study. In order to avoid the disappointment bias, they will be randomized into three groups, according to a procedure adapted from the Zelen method, in two stages. After verification of the inclusion criteria, eligible patients will receive initial information detailing the follow-up methods, but not the intervention. If patients agree to participate, they will be randomized to three groups: CAT, MBCT or usual management. Patients in the CAT and MBCT groups will then be informed of the group in which they have been randomized, will sign a new consent form and the corresponding intervention will be offered to them.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CAT (Experimental): induction of cognitive dissonance
  Interventions: Other: CAT
- MBCT (Experimental): TCA-specific mindfulness approach
  Interventions: Other: CAT
- TAU (No Intervention): usual support

INTERVENTIONS:
Other: CAT — 2 group programs, led by trained speakers, addressing specific ED topics through written, verbal and/or behavioral exercises,
  Other Names: MBCT
  Arms: CAT; MBCT

SUMMARY:
This study propose to compare the effectiveness of two care programs, the CAT and cognitive therapy based on mindfulness (Mindfulness-Based Cognitive Therapy, MBCT) compared to the usual care ("Treated as usual", TAU) in AM and to show their benefit on dimensions specific to EDs such as body dissatisfaction and the internalization of the ideal of thinness, but also on eating symptoms and the anxious and depressive dimensions.

DETAILED DESCRIPTION:
The patients will be recruited from the active files of the four centers participating in the study. In order to avoid the disappointment bias, they will be randomized into three groups, according to a procedure adapted from the Zelen method, in two stages. After verification of the inclusion criteria, eligible patients will receive initial information detailing the follow-up methods, but not the intervention. If patients agree to participate, they will be randomized to three groups: CAT, MBCT or usual management. Patients in the CAT and MBCT groups will then be informed of the group in which they have been randomized, will sign a new consent form and the corresponding intervention will be offered to them.

Experimental group: 2 group programs, led by trained facilitators, addressing specific ED topics through written, verbal and/or behavioral exercises,

* by following a directive standardized manual aimed at inducing cognitive dissonance (CAT group)
* via a specific TCA mindfulness approach (MBCT group) Control group: usual management (TAU). Same number of sessions as the experimental group (8 weekly sessions), consisting of supportive psychotherapy, +/- adjunctive drug treatment, symptomatic.

HibernAM ancillary study:

For patients with restrictive anorexia nervosa, serum collection on inclusion. Collection of serum from blood samples taken as part of routine care for matched healthy subjects.

Addition of serum from patients with restrictive anorexia nervosa, and from matched healthy subjects, to human myotubes in culture for the exploration of protein metabolism

ELIGIBILITY:
Inclusion Criteria:

* Anorexia nervosa as defined by the DSM-5 (anorexia nervosa of pure restrictive type F50.01 or purgative type F50.02),
* 14 < BMI < 18.5 (outpatient management possible)
* Affiliation to a social security scheme or beneficiary of such a scheme
* Signed informed consent

Exclusion Criteria:

* other group support of their TCA
* regular psychological follow-up for a main psychiatric disorder other than TCA
* mental retardation or psychiatric pathology other than TCA or severe somatic not allowing efficient participation in the therapeutic program and interviews
* presence, at the time of the study, of a chronic condition that typically affects weight (digestive disease such as celiac disease, Crohn's disease; malignant tumor pathology; endocrine pathology such as hypo/hyperthyroidism, hyper/ hypocortisolism, pituitary or hypothalamic tumor, etc.).
* refusal to participate in the study
* pregnant, lactating women
* period of exclusion from another study,
* administrative or judicial supervision
* subject cannot be contacted in case of emergency

Ancillary study: Volunteers will be excluded from the control group:

* having a significant biological abnormality
* a history of TCA or pathology likely to impact protein metabolism,
* pregnancy or breastfeeding at the time of the blood sample,
* under guardianship, deprivation of liberty, administrative or judicial supervision and exclusion from another study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Score of the Body Shape Questionnaire BSQ-34 self-administered questionnaires at 3 months, adjusted to the initial score (D0). | 3 months
  The main objective is to compare the effectiveness of CAT and MBCT programs compared to the usual care, on the reduction of body dissatisfaction, in patients presenting with AM. If one or both of these methods are superior to the usual support, we will compare them with each other following a hierarchical sequential analysis method.
  months, adjusted to the initial score (D0).
  The attitudinal dimension of body image can be assessed using the "Body Shape Questionnaire" (BSQ)-34, a one-dimensional self-questionnaire composed of 34 items assessing body dissatisfaction. (BSQ; Cooper, Taylor, Cooper, & Fairburn, 1986). A French version was validated in 2005 [68].
  Full BSQ score Classification less than 80= no concern with shape 80 to 110= mild concern with shape 111 to 140= moderate concern with shape over 140= marked concern with shape

CONTACTS AND LOCATIONS:
Overall Officials: Mircea Polosan, Principal Investigator — University Hospital, Grenoble
Locations (1):
- Julien Colombat, Grenoble, France